CLINICAL TRIAL: NCT05784389
Title: Reduction of Metabolic Acidosis in Patients With Chronic Kidney Disease in Stage 4 and 5
Acronym: REMA-CKD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-21069570
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Kidney Diseases; Metabolic Acidosis; Renal Insufficiency; CKD; Pre-dialysis
Keywords: Potential renal acid load; PRAL; Study design; Diet; Humans; Elderly; Bicarbonate/blood; Muscle strength; Hand strength; Chair stand test; Calorimetry, indirect; Bone mineralization; Carbon dioxide/blood; Phosphor/urine; Potassium/urine; Urea/blood; Urea/urine
MeSH Terms: conditions — Kidney Diseases; Acidosis; Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
  Crossover design: 1 arm consisting of three consecutive periods of two weeks (control, intervention and follow up).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low PRAL diet (Experimental): Experimental: Low PRAL diet Crossover design: 1 arm consisting of three consecutive periods of two weeks (control, intervention and follow up).
  Interventions: Other: Low PRAL

INTERVENTIONS:
Other: Low PRAL — Two weeks on a low PRAL diet compared to 2 week free living

SUMMARY:
This clinical trial aims to investigate and test the effect of an acid/base diet in chronic kidney disease (CKD) patients, CKD stage 4 and 5. The trial is guided by the hypothesis that an acid/base diet will reduce the degree of acidosis and simultaneously reduce the need for bicarbonate supplements.

DETAILED DESCRIPTION:
Observational studies indicate that diets with a low "potential renal acid load (PRAL)" is associated with a lower serum-bicarbonate value. Therefore, we aim to investigate this association through an interventional study design.

Participants will be asked to follow a restricted diet with a low "PRAL" during a 6-week trial divided into three periods: two-week of free-living control, two-weeks of intervention, and a two-week free-living follow-up.

The PRAL calculation tool will be used to create a diet low in acid and to develop individualized diet plans for each patient. The diet will comply with Danish national guidelines on threshold for potassium and protein, due to the high risk of hyperkalemia in CKD patients. The patients will be asked to document their food and drink intake by taking pictures of their plates and cups before and after a meal, over a 24-hour period.

ELIGIBILITY:
Inclusion Criteria:

* Chronic acidosis (plasma-bicarbonate under 22 mmol/l at multiple measures within the last 12 months).
* Diagnosed with non-dialysis needed chronic kidney disease in stage 4 and 5 (eGFR below 30 ml/min/1,73 m2)
* Of legal age and over 18 of years
* Understand danish and understand the written material
* Able to cooperate about the diet
* Able to take pictures with their phone or willing to learn

Exclusion Criteria:

* Vegan and vegetarian with very low intake of animal protein (below 25 g/day)
* Pregnant or breast feeding
* Patients with short bowel syndrome, bricker bladder, pancreatitis or any other known malabsorption problem
* Potassium above 5 mmol/l
* Ongoing infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
Plasma-total carbon dioxide (CO2) | 6 weeks
  mmol/l

SECONDARY OUTCOMES:
Plasma-alkaline phosphatase | 6 weeks
  U/l
Plasma-sodium ion | 6 weeks
  mmol/l
Plasma-creatinine | 6 weeks
  umol/l
Plasma-parathyroid hormone | 6 weeks
  pmol/l
Plasma-carbamide | 6 weeks
  mmol/l
Plasma-albumin | 6 weeks
  g/l
Urine-phosphorous | 6 weeks
  mmol/d
Urine-sodium | 6 weeks
  mmol/d
Urine-potassium | 6 weeks
  mmol/d
Urine-carbamide | 6 weeks
  mmol/d
Urine-albumin | 6 weeks
  mg/d
Urine-magnesium | 6 weeks
  mmol/d
Urine-creatinine | 6 weeks
  mmol/d
Urine-calcium | 6 weeks
  mmol/d
Total acid excretion in urine | 6 weeks
  mmol/d
Urine-pH | 6 weeks
  pH
Urine ammonium-ion (NH4+) excretion | 6 weeks
  mmol/d
Urine net acid excretion | 6 weeks
  mmol/d
Urine bicarbonate | 6 weeks
  mmol/l

OTHER OUTCOMES:
Plasma-Potassium | 6 weeks
  mmol/l
Plasma-calcium | 6 weeks
  mmol/l
Plasma-magnesium | 6 weeks
  mmol/l
Plasma-inorganic phosphorous | 6 weeks
  mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Lisbet Brandi, Doctor Med, Principal Investigator — Nordsjaellands Hospital; Jens R Andersen, As. prof., Principal Investigator — University of Copenhagen
Locations (1):
- Nordshjaellands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No
sharing is not currently possible recording to legislation and consent form.